CLINICAL TRIAL: NCT06519513
Title: 'The Effect of Laughter Yoga on Midwives' Perceived Stress Level and Burnout Level: Randomized Controlled Study'
Brief Title: Laughter Yoga, Stress Level and Burnout Level
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Asssociate professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KırklareliAS-11
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Burnout, Psychological; Stress; Laughter
Keywords: stress; burnout; laughter yoga
MeSH Terms: conditions — Burnout, Psychological; Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter yoga group (Experimental): Laughter yoga will be performed in 8 sessions, 2 days a week for 4 weeks. The duration of each session will be 40 minutes. Laughter yoga sessions will be held on a day suitable for all participants and with the participation of at least 8 people. The session will start with warm-up exercises and continue with laughter exercises. People in the group will do these exercises with the guidance of the researcher.
  Interventions: Other: Laughter yoga
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practice on their own to reduce stress and burnout levels. The researcher will ask the participants via phone 4 times a week for 1 month whether they have taken any action to reduce their stress and burnout symptoms. Participants who use any of the pharmacological or non-pharmacological practices to reduce stress and burnout symptoms will be excluded from the study.

INTERVENTIONS:
Other: Laughter yoga — Part 1: Deep Breathing Exercises: Raise the arms up towards the sky and take a deep breath as possible and hold the breath for 4-5 seconds. This application is repeated several times. This section takes approximately 5-10 minutes.
  Part 2: Warm-up exercises: Hands are kept parallel to each other and clapped. The tips of the fingers and palms touch each other, the acupuncture points on both hands are stimulated and the individual's energy level increases.
  Section 3: Childish Games: In this section there are childish games. These games are visualized in the mind and the participants are asked to raise their arms upwards in the shape of the letter "Y".This section takes approximately 10 minutes.
  Section 4: Laughter Exercises: Participants are given verbal guidance such as "Put your hand on your heart, feel your heartbeat, let's exhale with a smile, let's make a wish or pray" and the laughter exercise is terminated. This section takes approximately 15 minutes.
  Arms: Laughter yoga group

SUMMARY:
The positive interaction between personal and business life results in the health of the healthcare personnel and the success of the institution. Burnout, which occurs as a result of a crisis in an individual's working life, manifests itself as fatigue, lack of energy, feeling inadequate in the professional role and lack of confidence.

Laughter, which helps people to endure stressful situations or processes, improves a person's problem-solving ability by reducing depression and increasing insight. For this reason, laughter reduces a person's exposure to negative environmental cues and helps them with self-control. Laughter, a positive emotion, appears to be a useful and healthy way to cope with stress. The aim of the research to be conducted is to evaluate the effect of laughter yoga on the stress and burnout levels of midwives.

DETAILED DESCRIPTION:
The positive interaction between personal and business life results in the health of the healthcare personnel and the success of the institution.

People who are satisfied with their working environment work more efficiently. High job satisfaction levels of midwives who ensure that newborns, pregnant women and postpartum women, as well as newborns, pregnant women and postpartum mothers, receive quality care will ensure that the service they provide will be of higher quality.

Burnout, which occurs as a result of a crisis in an individual's working life, manifests itself as fatigue, lack of energy, feeling inadequate in the professional role and lack of confidence. This situation, which occurs in the healthcare worker, will negatively affect the quality of patient care as it will cause a regression in the healthcare worker's decision-making process and an increase in medical errors. Laughter, which helps people to endure stressful situations or processes, improves a person's problem-solving ability by reducing depression and increasing insight. For this reason, laughter reduces a person's exposure to negative environmental cues and helps them with self-control. Laughter, a positive emotion, appears to be a useful and healthy way to cope with stress. People gain a positive mood through laughter, and a negative mood, thought or personality can also be changed in a positive way. Laughter therapy, which is used to increase psychosocial behaviors, positively affects the general quality of life.

The aim of the research to be conducted is to evaluate the effect of laughter yoga on the stress and burnout levels of midwives.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Answering survey and scale forms fully
* Social media accounts, presence in WhatsApp groups
* Ability to read and understand Turkish
* 5 years or more of working life in the profession
* Not having any health problems that would prevent communication
* Working in a maternity ward or gynecology ward
* Scoring 14 or above on the perceived stress scale

Exclusion Criteria:

* Not volunteering to participate in the research
* Answering survey and scale forms incompletely
* Not understanding Turkish
* Less than 5 years of working life in the profession
* Having any health problem that prevents communication
* Working outside the maternity ward or gynecology ward

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Enrollment: 80 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Burnout Scale | between 2 to 4 weeks
  Developed by Pines and Aronson (1988) to be used on non-professional groups as well as all professional groups, the TOS consists of twenty-one items prepared as self-report on a seven-point scale to evaluate the physical, emotional and mental exhaustion level of individuals.
Perceived Stress Scale-10 | between 2 to 4 weeks
  It measures the extent to which situations in a person's life are evaluated as stressful. Scores of 0-13 are considered low stress. Scores between 14 and 26 are considered moderate stress. Scores between 27 and 40 are considered high perceived stress.

SECONDARY OUTCOMES:
General Health Survey-28 | between 2 to 4 weeks
  It is a screening test created by the individual to detect mental health problems encountered in society and non-psychiatric clinical environments. A minimum of 0 and a maximum of 28 points can be obtained from the scale. A higher total score increases the likelihood of psychological problems.

CONTACTS AND LOCATIONS:
Overall Officials: AYCA SOLT KIRCA, Phd, Study Chair — Kırklareli University
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided